CLINICAL TRIAL: NCT00816296
Title: Evaluation of the Intestinal Microbiome in Obese Children With and Without Non-Alcoholic Fatty Liver Disease
Brief Title: Evaluation of Intestinal Microbiome in Obese Kids
Status: Withdrawn | Type: Observational
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Vincent Biank, Medical College of Wisconsin
Other Study IDs: CHW 08/159; GC 727
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Obesity; Microbiome
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will need to give a blood and stool samples on 3 separate occasions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Obese (BMI>30) and normal AST and ALT. Between the ages of 5 and 18 years old.
  Interventions: Other: Blood Draw; Other: Stool collection; Other: BodPod Measurement; Other: Liver Ultrasound
- Liver Disease: Obese (BMI>30) and elevated AST and/or ALT (evidence of NAFLD). Between the ages of 5 and 18 years old.
  Interventions: Other: Blood Draw; Other: Stool collection; Other: BodPod Measurement; Other: Liver Ultrasound

INTERVENTIONS:
Other: Blood Draw — 2 tablespoons of blood will be drawn from participants at study entry, 3 months after study entry, and 6 months after study entry.
Other: Stool collection — Stool will be collected from participants 3 times during the study -- at study entry, 3 months from study entry, and 6 months after study entry.
Other: BodPod Measurement — Body composition will be measured using a BodPod at study entry, 3 months after study entry, and 6 months after study entry.
Other: Liver Ultrasound — A liver ultrasound will be performed at study entry and 6 months after study entry.

SUMMARY:
The goal of this study is to investigate comparisons between the intestinal microbiome in patients with obesity and in patients with obesity and Non-Alcoholic Fatty Liver Disease (NAFLD). With this protocol we hope to better understand how the microbiome of each individual works with disease progression.

DETAILED DESCRIPTION:
The goal of this study is to investigate and compare the composition of the intestinal microbiome in patients with obesity only to patients with obesity and Non-Alcoholic Fatty Liver Disease (NAFLD). In addition, we will investigate the relationship between alterations in the intestinal microbiome, immune activation, and the progression of NAFLD to Non-Alcoholic Steatohepatitis (NASH). We hypothesize that alterations in the intestinal microbiome are associated with increased immune activation and progression of obesity associated NAFLD. Based on this hypothesis we propose the following aims:

Aim 1. Identify and enroll pediatric cohort with obesity or obesity/NAFLD to study the role of the intestinal microbiome on the development of NAFLD.

1. Enroll participants through the NEW Kids program for treatment of pediatric obesity at Children's Hospital of Wisconsin (CHW). Identify and classify participants through initial clinical evaluation, collect clinical metadata, and obtain and process blood and stool samples for analysis. Demonstrate feasibility by showing that participants can be recruited and participate in the specific study protocol.
2. Follow study population through nutritional/exercise intervention, with follow up collection of clinical data, stool, and blood samples.

Aim 2. Characterize the intestinal microbiome through quantitative PCR and high throughput sequencing analysis of stool specimens in participants with obesity and obesity/NAFLD.

1. Demonstrate feasibility by showing that sampling aliquots from patient fecal samples can be successfully analyzed by proposed methods and yield consistent results for duplicate samples.
2. Compare sequencing results and metagenomic analysis for study groups with particular attention to bacterial composition and metabolic capacity associated with energy harvest, lipid and carbohydrate transport, enhancement of epithelial barrier integrity, and choline metabolism.
3. Investigate whether intervention (nutritional/exercise) results in longitudinal alterations in the intestinal microbiome.

Aim 3. Characterize evidence of systemic inflammation by C-reactive protein (CRP), Tumor necrosis factor alpha (TNF-alpha)Transforming growth factor beta 1 (TGF-beta and LPS Binding Protein (LBP) levels, and analyze results in relationship to the intestinal microbiome and the presence of NAFLD.

1. Compare levels of systemic inflammatory markers of participants with obesity vs. obesity/NAFLD
2. Investigate whether intervention (nutritional/exercise) results in longitudinal alterations in systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18 Years old
* Willing to consent/undergo necessary procedures
* Obese (BMI>30)
* Speak English or Spanish

Exclusion Criteria:

* any other causes of liver disease
* any chronic illnesses or life threatening conditions

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Gastroenterology Clinic at Children's Hospital of Wisconsin
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Alterations in the intestinal microbiome are associated with increased immune activation and progression of obesity associated NAFLD. | 3 years

SECONDARY OUTCOMES:
Characterize the intestinal microbiome through quantitative analysis of stool samples in participants with obesity and those with obesity and NAFLD. | 3 years
Characterize inflammatory markers of participants with obesity versus those obese participants that also have NAFLD. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Biank, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Angulo P, Keach JC, Batts KP, Lindor KD. Independent predictors of liver fibrosis in patients with nonalcoholic steatohepatitis. Hepatology. 1999 Dec;30(6):1356-62. doi: 10.1002/hep.510300604. PMID 10573511
- [Background] Iacobellis A, Marcellini M, Andriulli A, Perri F, Leandro G, Devito R, Nobili V. Non invasive evaluation of liver fibrosis in paediatric patients with nonalcoholic steatohepatitis. World J Gastroenterol. 2006 Dec 28;12(48):7821-5. doi: 10.3748/wjg.v12.i48.7821. PMID 17203527
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Li Z, Soloski MJ, Diehl AM. Dietary factors alter hepatic innate immune system in mice with nonalcoholic fatty liver disease. Hepatology. 2005 Oct;42(4):880-5. doi: 10.1002/hep.20826. PMID 16175608
- [Background] Brun P, Castagliuolo I, Di Leo V, Buda A, Pinzani M, Palu G, Martines D. Increased intestinal permeability in obese mice: new evidence in the pathogenesis of nonalcoholic steatohepatitis. Am J Physiol Gastrointest Liver Physiol. 2007 Feb;292(2):G518-25. doi: 10.1152/ajpgi.00024.2006. Epub 2006 Oct 5. PMID 17023554
- [Background] Fields DA, Goran MI, McCrory MA. Body-composition assessment via air-displacement plethysmography in adults and children: a review. Am J Clin Nutr. 2002 Mar;75(3):453-67. doi: 10.1093/ajcn/75.3.453. PMID 11864850
- [Background] Nicholson JC, McDuffie JR, Bonat SH, Russell DL, Boyce KA, McCann S, Michael M, Sebring NG, Reynolds JC, Yanovski JA. Estimation of body fatness by air displacement plethysmography in African American and white children. Pediatr Res. 2001 Oct;50(4):467-73. doi: 10.1203/00006450-200110000-00008. PMID 11568289